CLINICAL TRIAL: NCT00084084
Title: An Open Label Clinical Trial of Replagal Enzyme Replacement Therapy In Children With Fabry Disease Who Have Completed Study TKT023 or Who Are Naive to Enzyme Replacement Therapy
Brief Title: Replagal Enzyme Replacement Therapy for Children With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKT029
Record Dates: First submitted 2004-06-05; First posted 2004-06-07 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Fabry Disease
Keywords: Lysosomes; Storage; Glycolipid; Fabry disease; Stroke; Children; Pediatrics
MeSH Terms: conditions — Fabry Disease; Stroke | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Agalsidase alfa (Cohort 1) (Experimental): Cohort 1: Patients who completed TKT023.
  Interventions: Drug: Agalsidase alfa
- Agalsidase Alfa (Cohort 2) (Experimental): Cohort 2: Treatment-naive patients.
  Interventions: Drug: Agalsidase alfa

INTERVENTIONS:
Drug: Agalsidase alfa — 0.2 mg/kg agalsidase alfa administered by IV infusion over 40 (+/- 10) minutes every other week for 52 weeks, with periodic reassessments for study continuation beyond 52 weeks
  Other Names: Replagal

SUMMARY:
Primary Objective(s):

* To assess the safety of Replagal at a dose of 0.2 mg/kg administered over 40 (+/-10) minutes in children with Fabry disease
* To assess the effect of Replagal on heart rate variability in patients 7 to 17 years of age

Secondary Objective(s):

* To determine the pharmacokinetics of Replagal at baseline and after the initiation of enzyme replacement therapy (ERT)
* To determine exploratory measurements of efficacy including renal function (ie, estimated glomerular filtration rate [eGFR] and creatinine clearance), clinical outcomes (in Cohorts 1 and 2), and sweating and left ventricular mass index (LVMI) (Cohort 1, Phase 1 only)

DETAILED DESCRIPTION:
TKT029 is an open label multi-center study to assess the safety of enzyme replacement therapy with Replagal (agalsidase alfa) in children with Fabry disease, who have completed 6 months of agalsidase alfa therapy in study TKT023 (Cohort 1) or who are treatment-naïve (Cohort 2) and meet all inclusion/exclusion criteria of this study. The study will consist of every other week treatment with Replagal for 52 weeks, with periodic reassessments by Shire HGT for continuation of the study beyond 52 weeks. A decision on the part of the study sponsor to terminate the study may be made at any time.

In Cohort 1, safety and clinical measurement assessments performed during Week 25 or 26 of Study TKT023 served as the baseline assessments for TKT029. Patients in Cohort 1 began treatment with Replagal manufactured using a roller bottle process (Replagal RB); this portion of treatment is denoted as Cohort 1, Phase 1. Safety evaluation visits for Cohort 1, Phase 1 were to be performed at Weeks 13, 25, 55, and every 26 weeks thereafter until the patient discontinued from the study or transitioned to treatment with Replagal manufactured using a bioreactor process (Replagal AF). The transition to Replagal AF marked the restart of the study clock and was denoted as Cohort 1, Phase 2. Safety evaluation visits for Cohort 1, Phase 2 will be performed at Weeks 1, 13, 25, 55, and every 26 weeks thereafter until the patient discontinues from or the sponsor terminates the study.

Patients in Cohort 2 will receive treatment with Replagal AF only; therefore there is only 1 study phase for these patients. Screening assessments performed at Week -1 will serve as the baseline assessments for this study. Safety evaluation visits for Cohort 2 will be performed at Weeks 13, 25, 37, 55 and every 26 weeks thereafter until the patients discontinues from or the sponsor terminates the study.

The final study visit for both cohorts will follow 30 days after the study study drug infusion, at which time a final safety evaluation will be performed. Patients who complete the study will be interviewed by telephone 30 days after their last study infusion for resolution of any outstanding adverse events (AEs) or concomitant medication changes. Any patient who withdraws early from the study will have a final study visit 30 days after the last study drug infusion, at which time a final safety evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

1a. For Cohort 1 (both phases):

- Patients must have completed all study requirements and assessments for Study TKT023 less than 30 (+/-7) days prior to enrolling in Study TKT029 and must have no safety or medical issues that contraindicate participation.

OR

1b. For Cohort 2:

* The patient is between 7 and 17 years of age at the time of informed consent, inclusive.
* The patient must be ERT-naive.
* The patient is a hemizygous male with Fabry disease as confirmed by a deficiency of alpha-galactosidase A activity measured in serum, leukocytes, or fibroblasts. Male patients who do not already have a documented deficiency of alpha-galactosidase A activity will provide a blood sample during screening for determination of alpha-galactosidase A activity level in their serum.

OR

- The patient is a heterozygous female or hemizygous male with Fabry disease as confirmed by a mutation of the alpha-galactosidase A gene. Patients who do not already have a documented mutation of the alpha-galactosidase A gene will provide a blood sample during screening for genotyping.

2. Adequate general health (as determined by the Investigators) to undergo the specified phlebotomy regimen and protocol-related procedures and no safety or medical contraindications for participation.

3. The minor child must assent to participate in the protocol and the parent(s) or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved informed concent form after all relevant aspects of the study have been explained and discussed with the child and the child's parent(s) or legal guardian(s).

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this study:

* Patient and/or the patient's parent(s) or legal guardian(s) are unable to understand the nature, scope, and possible consequences of the study.
* Patient is unable to comply with the protocol, e.g., uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for safety evaluations, or is otherwise unlikely to complete the study, as determined by the Investigator or the medical monitor.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2004-06-10 (Actual); Primary Completion 2011-06-15 (Actual); Study Completion 2011-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- United States (13):
  - Tucson Access Center of Arizona Kidney Disease Hypertension Center, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Children's Physician Group, Palm Beach Gardens, Florida
  - Christus St. Patrick Hospital, Lake Charles, Louisiana
  - Clinical Center, National Institutes of Health, Bethesda, Maryland
  - Memorial Hospital, Easton, Maryland
  - St. Louis Children's Hospital, St Louis, Missouri
  - NYU School of Medicine, New York, New York
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - University of Tennessee, Health Science Center, Memphis, Tennessee
  - Institute of Metabolic Diseases, Dallas, Texas
  - Office of Michael Cohen, Stafford, Virginia
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Schiffmann R, Pastores GM, Lien YH, Castaneda V, Chang P, Martin R, Wijatyk A. Agalsidase alfa in pediatric patients with Fabry disease: a 6.5-year open-label follow-up study. Orphanet J Rare Dis. 2014 Nov 26;9:169. doi: 10.1186/s13023-014-0169-6. PMID 25425121

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patient was enrolled in Cohort 2 (ie, no treatment-naive patients were enrolled).
Groups:
- Agalsidase Alfa (Cohort 1): Cohort 1 was composed of patients who had completed TKT023. Patients received 0.2 mg/kg agalsidase alfa, IV, every other week.
Period: Phase 1 (Treatment With Replagal RB)
Arm/Group | Agalsidase Alfa (Cohort 1)
Started | 17
Completed | 16
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Phase 2 (Transition to Replagal AF)
Arm/Group | Agalsidase Alfa (Cohort 1)
Started | 11 (The 11 patients remaining in TKT029 at the time Replagal AF was made available continued to Phase 2.)
Completed | 10
Not Completed | 1
Not completed — Failure to visit clinic as scheduled | 1

BASELINE CHARACTERISTICS:
Groups:
- Agalsidase Alfa (Cohort 1): 0.2 mg/kg agalsidase alfa infused by IV over 40 (+/- 10) minutes every other week
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.99 (3.2464)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15
  Hispanic | 2
Baseline Heart Rate Variability (SDNN) [Mean (Standard Deviation); unit: msec] — SDNN is defined as the standard deviation of all filtered RR intervals over the length of the analysis.
  msec | 98.947 (32.324)

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Experienced At Least One Adverse Event (AE)
Time Frame: 362 weeks
Population: Safety Population: Patients in Cohort 1 who received at least one dose of Replagal RB in Phase 1.
Measure: Number; unit: participants
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 17
participants | 17

2. Secondary Outcome: Pharmacokinetics - Area Under the Serum Concentration-Time Curve (AUC0-∞) - Week 81
Description: AUC0-∞ is a measure of the total exposure to a drug.
Time Frame: Pre-infusion; and post-infusion at 20, 40, 50, 60, 90 minutes, and 2, 3, 4, 8 hours.
Population: PK Population: All patients who received at least 1 dose of Replagal (RB or AF) and had at least 1 PK sample drawn.
Measure: Mean (Standard Deviation); unit: min·U/mL
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 11
min·U/mL | 245282 (159071)

3. Secondary Outcome: Pharmacokinetics - Area Under the Serum Concentration-Time Curve (AUC0-∞) - Week 133
Description: AUC0-∞ is a measure of the total exposure to a drug.
Time Frame: Pre-infusion; and post-infusion at 20, 40, 50, 60, 90 minutes, and 2, 3, 4, 8 hours.
Population: PK Population: All patients who received at least 1 dose of Replagal (RB or AF) and had at least 1 PK sample drawn.
Measure: Mean (Standard Deviation); unit: min·U/mL
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 11
min·U/mL | 295779 (161058)

4. Secondary Outcome: Pharmacokinetics - Area Under the Serum Concentration-Time Curve (AUC0-∞) - Week 159
Description: AUC0-∞ is a measure of the total exposure to a drug.
Time Frame: Pre-infusion; and post-infusion at 20, 40, 50, 60, 90 minutes, and 2, 3, 4, 8 hours.
Population: PK Population: All patients who received at least 1 dose of Replagal (RB or AF) and had at least 1 PK sample drawn.
Measure: Mean (Standard Deviation); unit: min·U/mL
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 11
min·U/mL | 218078 (73560)

5. Secondary Outcome: Pharmacokinetics - Area Under the Serum Concentration-Time Curve (AUC0-∞) - Week 315/341
Description: AUC0-∞ is a measure of the total exposure to a drug.
Time Frame: Pre-infusion; and post-infusion at 20, 40, 50, 60, 90 minutes, and 2, 3, 4, 8 hours.
Population: PK Population: All patients who received at least 1 dose of Replagal (RB or AF) and had at least 1 PK sample drawn.
Measure: Mean (Standard Deviation); unit: min·U/mL
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 11
min·U/mL | 213193 (119581)

6. Other Pre Specified Outcome: Heart Rate Variability - Change From Baseline at Week 185 in SDNN
Description: Heart rate variability was assessed by 2-hour Holter monitoring. Standard deviation of all filtered RR intervals over the length of the analysis (SDNN) was measured.
Time Frame: Week 185
Population: Number of participants present at Visit Week 185 included for analysis.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 9
msec | 20.256 (29.060)

7. Secondary Outcome: Pharmacokinetics - Maximum Observed Serum Concentration (Cmax) - Week 81
Description: Cmax is the peak plasma concentration of a drug after administration.
Time Frame: Pre-infusion; and post-infusion at 20, 40, 50, 60, 90 minutes, and 2, 3, 4, 8 hours.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 11
U/mL | 3173 (969)

8. Secondary Outcome: Pharmacokinetics - Maximum Observed Serum Concentration (Cmax) - Week 133
Description: Cmax is the peak plasma concentration of a drug after administration.
Time Frame: Pre-infusion; and post-infusion at 20, 40, 50, 60, 90 minutes, and 2, 3, 4, 8 hours.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 11
U/mL | 3842 (1235)

9. Secondary Outcome: Pharmacokinetics - Maximum Observed Serum Concentration (Cmax) - Week 159
Description: Cmax is the peak plasma concentration of a drug after administration.
Time Frame: Pre-infusion; and post-infusion at 20, 40, 50, 60, 90 minutes, and 2, 3, 4, 8 hours.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 11
U/mL | 3842 (1235)

10. Secondary Outcome: Pharmacokinetics - Maximum Observed Serum Concentration (Cmax) - Week 315/341
Description: Cmax is the peak plasma concentration of a drug after administration.
Time Frame: Pre-infusion; and post-infusion at 20, 40, 50, 60, 90 minutes, and 2, 3, 4, 8 hours.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Agalsidase Alfa (Cohort 1)
Number analyzed (Participants) | 11
U/mL | 3568 (1492)

ADVERSE EVENTS:
Time Frame: 362 weeks
Groups:
- Safety Population RB: Patients in Cohort 1 who received at least 1 dose of Replagal RB in Phase 1 - no data from Phase 2 (Replagal AF) included.
- Transition Safety Population: A subset of patients from the Safety Population RB who additionally received at least 1 dose of Replagal AF in Phase 2.
Arm/Group | Safety Population RB | Transition Safety Population
Serious Adverse Events (participants affected / at risk) | 2/17 | 2/11
Other Adverse Events (participants affected / at risk) | 17/17 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population RB (N=17) | Transition Safety Population (N=11)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (2) | 1 (2)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Renal Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pectus Excavatum (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population RB (N=17) | Transition Safety Population (N=11)
Gastroenteritis Viral (Infections and infestations) | 8 (12) | 5 (6)
Nasopharyngitis (Infections and infestations) | 7 (12) | 6 (12)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (11) | 5 (16)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Ear Infection (Infections and infestations) | 2 (3) | 2 (3)
Sinusitis (Infections and infestations) | 2 (5) | 4 (8)
Acarodermatitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 1 (2)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 1 (1)
Infected Bites (Infections and infestations) | 1 (1) | 1 (1)
Infectious Mononucleosis (Infections and infestations) | 1 (1) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 1 (2) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Rocky Mountain Spotted Fever (Infections and infestations) | 1 (1) | 1 (1)
Tinea Pedis (Infections and infestations) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Blister Infected (Infections and infestations) | 0 (0) | 1 (1)
Body Tinea (Infections and infestations) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 0 (0) | 1 (1)
Molluscum Contagiosum (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Attention Deficit / Hyperactivity Disorder (Psychiatric disorders) | 3 (4) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (2)
Decreased Activity (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (3)
Panic Disorder (Psychiatric disorders) | 1 (2) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 9 (33) | 7 (46)
Neuralgia (Nervous system disorders) | 9 (35) | 7 (32)
Burning Sensation (Nervous system disorders) | 6 (16) | 5 (15)
Paraesthesia (Nervous system disorders) | 3 (7) | 3 (7)
Balance Disorder (Nervous system disorders) | 2 (2) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (5) | 1 (5)
Coordination Abnormal (Nervous system disorders) | 1 (1) | 1 (1)
Cranial Nerve Disorder (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Facial Paresis (Nervous system disorders) | 1 (3) | 1 (3)
Hypersomnia (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Poor Quality Sleep (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Reflexes Abnormal (Nervous system disorders) | 1 (3) | 1 (3)
Sinus Headache (Nervous system disorders) | 2 (2) | 1 (1)
Thalamic Infarction (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in Attention (Nervous system disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Eye Pain (Eye disorders) | 1 (2) | 1 (2)
Eye Swelling (Eye disorders) | 1 (1) | 1 (1)
Gaze Palsy (Eye disorders) | 1 (1) | 1 (1)
Myopia (Eye disorders) | 1 (2) | 1 (2)
Strabismus (Eye disorders) | 1 (1) | 1 (1)
Refraction Disorder (Eye disorders) | 0 (0) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 4 (6) | 1 (1)
Cerumen Impaction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Deafness Unilateral (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Middle Ear Effusion (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Arrhythmia Supraventricular (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (3)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 2 (6)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Pallor (Vascular disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (27) | 10 (23)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 10 (16) | 6 (14)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 5 (14)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (10)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 8 (13) | 8 (14)
Nausea (Gastrointestinal disorders) | 7 (11) | 5 (15)
Abdominal Pain Upper (Gastrointestinal disorders) | 6 (10) | 6 (12)
Vomiting (Gastrointestinal disorders) | 6 (13) | 6 (12)
Diarrhoea (Gastrointestinal disorders) | 4 (11) | 6 (17)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 3 (3)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2)
Aphthous Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal Incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Frequent Bowel Movements (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 1 (2) | 1 (3)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (6)
Erythema (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (5)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Angiokeratoma (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (5)
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (5) | 1 (6)
Vasculitic Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (9)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8 (59) | 8 (67)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 2 (9)
Groin Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Posture Abnormal (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Urethral Meatus Stenosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Testicular Pain (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Balanitis (Reproductive system and breast disorders) | 1 (2) | 1 (2)
Scrotal Pain (Reproductive system and breast disorders) | 1 (2) | 1 (2)
Testicular Oedema (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pectus Excavatum (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 12 (27) | 9 (19)
Chest Pain (General disorders) | 6 (9) | 7 (13)
Fatigue (General disorders) | 4 (5) | 4 (6)
Pain (General disorders) | 3 (5) | 4 (8)
Gait Disturbance (General disorders) | 2 (3) | 2 (4)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 5 (7)
Oedema Peripheral (General disorders) | 2 (2) | 2 (3)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest Discomfort (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Infusion Site Pain (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 1 (1)
Temperature Intolerance (General disorders) | 1 (1) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 2 (2)
Albumin Urine Present (Investigations) | 1 (1) | 0 (0)
Blood Albumin Increased (Investigations) | 1 (1) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1) | 1 (1)
Blood Triglycerides Increased (Investigations) | 1 (1) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1) | 1 (1)
Nuclear Magnetic Resonance Imaging Brain Abnormal (Investigations) | 1 (1) | 1 (1)
Pulmonary Function Test Decreased (Investigations) | 1 (1) | 1 (1)
Sputum Abnormal (Investigations) | 1 (1) | 1 (1)
Weight Decreased (Investigations) | 1 (2) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 5 (15) | 5 (16)
Excoriation (Injury, poisoning and procedural complications) | 5 (16) | 5 (16)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 4 (5) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 3 (8) | 3 (8)
Skin Laceration (Injury, poisoning and procedural complications) | 3 (9) | 3 (10)
Joint Injury (Injury, poisoning and procedural complications) | 2 (3) | 2 (3)
Joint Sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 2 (4) | 2 (4)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (3)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Heat Exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Renal Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (2) | 1 (2)
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤ 180 days from the time submitted to Shire for review. Shire does not prohibit publication but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.